CLINICAL TRIAL: NCT04254900
Title: Energy Availability in Wheelchair Athletes
Brief Title: Energy Availability in Male and Female Elite Wheelchair Athletes Over Seven Consecutive Training Days
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2018-35
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Energy Supply; Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male wheelchair athletes: Other
  Interventions: Other: evaluating energy availability
- Female wheelchair athletes: Other
  Interventions: Other: evaluating energy availability

INTERVENTIONS:
Other: evaluating energy availability — energy availability will be determined by measuring energy intake, exercise energy expenditure and fat-free mass and using the following formula: energy availability = (energy intake - exercise energy expenditure) / fat-free mass

SUMMARY:
Low energy availability (LEA) is a major problem in sports as athletes ingest often a lower amount of energy compared to their actual needs. The availability of energy is calculated based on their daily energy intake and the energy cost of the daily training sessions in relation to their fat-free mass. Based on this calculation, it is known how much energy will available for the body (beside the fuel for training) to keep it in optimal physiological functioning. It has been shown, that LEA occurs very often in female athletes, in endurance athletes as well as athletes in weight-sensitive sports (i.e. jockeys, combat sports, gymnastics, ballet). The purpose of this study was to investigate, whether LEA is a problem in wheelchair athletes as well.

DETAILED DESCRIPTION:
Energy availability will be assessed over 7 consecutive training days using a dietary and training record as well as the Leisure Time PHysical Activity Questionnaire for spinal cord injury. Resting Energy expenditure will be measured as well as body composition (by a DXA) before the start of data collection.

ELIGIBILITY:
Inclusion Criteria:

* athletes from a national team in wheelchair sports

Exclusion Criteria:

* unable to follow normal training routine
* unable to record diet or training

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Elite wheelchair athletes from national team in different wheelchair sports
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
energy availability | 7 consecutive days during pre-season
  energy availability = (energy intake - exercise energy expenditure) / fat-free mass. Energy intake and exercise energy expenditure are measured using a food and training diary. The fat-free mass will be measured using a DXA scan.

CONTACTS AND LOCATIONS:
Overall Officials: Joelle Flueck, PhD, Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No